CLINICAL TRIAL: NCT03020160
Title: A Multicenter, Open-Label, Phase III Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Emicizumab Given Every 4 Weeks (Q4W) in Patients With Hemophilia A
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Emicizumab Given Every 4 Weeks in Participants With Hemophilia A
Acronym: HAVEN 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BO39182; 2016-001094-33 (EudraCT Number)
Record Dates: First submitted 2016-12-21; First posted 2017-01-13 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emicizumab: PK Run-in Cohort (Experimental): Participants received emicizumab subcutaneously (SC) at a dose of 6 mg/kg once every 4 weeks, with no loading dose, for at least 24 weeks.
  Interventions: Drug: Emicizumab
- Emicizumab: Expansion Cohort (Experimental): Participants received emicizumab subcutaneously (SC) at a loading dose of 3 mg/kg once every week for the first 4 weeks followed by a maintenance dose of 6 mg/kg emicizumab SC once every 4 weeks for at least 24 weeks.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Emicizumab will be administered according to dose and schedule described in respective arms. After at least 24 weeks on prophylactic emicizumab, individuals who experienced suboptimal bleeding control on emicizumab (according to protocol-defined criteria) had the opportunity to increase their dose to 3 mg/kg weekly. Upon implementation of protocol Version 5 (20-Dec-2019), treatment duration was extended. During this study prolongation, participants had the opportunity to switch to a preferred emicizumab dosing regimen (1.5 mg/kg weekly, 3 mg/kg every 2 weeks, or 6 mg/kg every 4 weeks) in order to provide them the same flexibility as with commercial product.
  Other Names: Hemlibra; RO5534262; ACE910

SUMMARY:
This multicenter, open-label, non-randomized study will assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of emicizumab administered at a dose of 6 milligrams per kilogram (mg/kg) every 4 weeks in participants with hemophilia A with or without inhibitors against factor VIII (FVIII). The study consists of 2 parts: a pharmacokinetic (PK) run-in part followed by an expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than or equal to (>/=) 40 kilograms (kg) at screening
* Diagnosis of severe congenital hemophilia A or hemophilia A with FVIII inhibitors
* Participants using rFVIIa or willing to switch to recombinant activated factor VII (rFVIIa) as primary bypassing agent for the treatment of breakthrough bleeds
* FVIII inhibitor test during screening with titer results available prior to first administration of study drug
* Participants without FVIII inhibitors, that is with less than (<) 0.6 Bethesda unit per milliliter [BU/mL];< 1.0 BU/mL only for laboratories with an historical sensitivity cutoff for inhibitor detection of 1.0 BU/mL, who completed successful immune tolerance induction (ITI) must have done so at least 5 years before screening and must have no evidence of inhibitor recurrence (permanent or temporary) indicated by detection of an inhibitor greater than (>) 0.6 BU/mL (> 1.0 BU/mL only for laboratories with an historical sensitivity cutoff for inhibitor detection of 1.0 BU/mL) since ITI
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than hemophilia A
* Ongoing or planned ITI therapy; participants in whom ITI has failed will be eligible with a 72-hour washout period prior to the first emicizumab administration
* History of illicit drug or alcohol abuse within 48 weeks prior to screening, in the investigator's judgment
* Participants who are at high risk for thrombotic microangiopathy (TMA) (for example, have a previous medical or family history of TMA), in the investigator's judgment
* Previous (within the last 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Other conditions (for example, certain autoimmune diseases) that may currently increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Known HIV infection with cluster of differentiation (CD) 4 cells counts <200 cells per microliter (cells/mcL)
* Use of systemic immunomodulators (for example, interferon) at enrollment or planned use during the study, with the exception of anti-retroviral therapy
* Concomitant disease, condition, significant abnormality on screening evaluations or laboratory tests, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an additional unacceptable risk in administering study drug to the participant
* Pregnancy or lactation or intention to become pregnant during the study
* Women with a positive serum pregnancy test result within 7 days prior to initiation of study drug

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (4):
  - University of California Davis, Sacramento, California
  - Indiana Hemophilia & Thrombosis center, Indianapolis, Indiana
  - University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Univ of N Carolina Chapel Hill; Hematology/Oncology, Chapel Hill, North Carolina
- Australia (2):
  - Royal Brisbane Hospital; Clinical Haematology, Brisbane, Queensland
  - Royal Adelaide Hospital; Haematology Clinical Trials, Adelaide, South Australia
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Japan (4):
  - Hokkaido University Hospital, Hokkaido
  - Nara Medical University Hospital, Nara
  - National Center for Child Health and Development, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Poland (2):
  - Instytut Hematologii i Transfuzjologii; Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw
  - Uniwersytecki Szpital Kliniczny; Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku, Wroclaw
- Spain (3):
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia

REFERENCES:
- [Derived] Kruse-Jarres R, Peyvandi F, Oldenburg J, Chang T, Chebon S, Doral MY, Croteau SE, Lambert T, Kempton CL, Pipe SW, Ko RH, Trzaskoma B, Dhalluin C, Bienz NS, Niggli M, Lehle M, Paz-Priel I, Young G, Jimenez-Yuste V. Surgical outcomes in people with hemophilia A taking emicizumab prophylaxis: experience from the HAVEN 1-4 studies. Blood Adv. 2022 Dec 27;6(24):6140-6150. doi: 10.1182/bloodadvances.2022007458. PMID 35939785
- [Derived] Pipe SW, Shima M, Lehle M, Shapiro A, Chebon S, Fukutake K, Key NS, Portron A, Schmitt C, Podolak-Dawidziak M, Selak Bienz N, Hermans C, Campinha-Bacote A, Kiialainen A, Peerlinck K, Levy GG, Jimenez-Yuste V. Efficacy, safety, and pharmacokinetics of emicizumab prophylaxis given every 4 weeks in people with haemophilia A (HAVEN 4): a multicentre, open-label, non-randomised phase 3 study. Lancet Haematol. 2019 Jun;6(6):e295-e305. doi: 10.1016/S2352-3026(19)30054-7. Epub 2019 Apr 16. PMID 31003963

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 7 patients were screened and enrolled in the PK run-in cohort of the study. For the expansion cohort, a total of 44 patients were screened, 41 of whom were enrolled.
Groups:
- Emicizumab: PK Run-In Cohort: Participants received emicizumab subcutaneously (SC) at a dose of 6 mg/kg once every 4 weeks (Q4W), with no loading dose, for at least 24 weeks. Upon implementation of protocol version 5 (20-Dec-2019), each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted (i.e., emicizumab SC 1.5 mg/kg once every week [QW], 3 mg/kg once every 2 weeks [Q2W], or 6 mg/kg Q4W) and continue on that dosing regimen until discontinuation from the study.
- Emicizumab: Expansion Cohort: Participants received emicizumab subcutaneously (SC) at a loading dose of 3 mg/kg once every week for the first 4 weeks followed by a maintenance dose of 6 mg/kg emicizumab SC once every 4 weeks (Q4W) for at least 24 weeks. Upon implementation of protocol version 5 (20-Dec-2019), each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted (i.e., emicizumab SC 1.5 mg/kg once every week [QW], 3 mg/kg once every 2 weeks [Q2W], or 6 mg/kg Q4W) and continue on that dosing regimen until discontinuation from the study.
Period: Overall Study
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Started | 7 | 41
Completed 24 Weeks in the Study | 7 | 41
Emicizumab Dose Was Up-Titrated | 0 | 4
Opted for a Change in Emicizumab Dosing Regimen (Upon Implementation of Protocol Version 5) | 0 | 1
Completed | 6 | 41
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort | Total
Number analyzed (Participants) | 7 | 41 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 4
  Between 18 and 65 years | 6 | 35 | 41
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 41 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 38 | 44
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 8 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 31 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Number of Participants with 0, 1, or >1 Target Joints in the Last 24 Weeks Prior to Study Entry [Count of Participants; unit: Participants] — A target joint was defined as a a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry.
  Participants
    0 Target Joints | 1 | 16 | 17
    1 Target Joint | 2 | 8 | 10
    >1 Target Joints | 4 | 17 | 21
Number of Participants by Hemophilia A Severity at Baseline [Count of Participants; unit: Participants]
  Mild | 0 | 1 | 1
  Moderate | 0 | 0 | 0
  Severe | 7 | 40 | 47
Number of Participants by Factor VIII Inhibitor Status at Baseline [Count of Participants; unit: Participants]
  Factor VIII Inhibitor Positive | 3 | 5 | 8
  Factor VIII Inhibitor Negative | 4 | 36 | 40

OUTCOME MEASURES:

1. Primary Outcome: Expansion Part: Annualized Bleeding Rate (ABR) for Treated Bleeds
Description: The number of treated bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and the first treatment thereafter and before a new bleed starts, are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to at least 24 weeks
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
treated bleed rate per year | 2.4 [1.38 to 4.28]

2. Primary Outcome: Expansion Part: Annualized Bleeding Rate (ABR) for All Bleeds
Description: The number of all bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: From Baseline to at least 24 weeks
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
all bleed rate per year | 4.5 [3.10 to 6.60]

3. Primary Outcome: Expansion Part: Annualized Bleeding Rate (ABR) for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A bleed is classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "treated spontaneous bleed" is a spontaneous bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Treated bleeds that fulfilled the 72-hour rule were included in the analysis of spontaneous bleeds. Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to at least 24 weeks
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Number (95% Confidence Interval); unit: treated spontaneous bleed rate per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
treated spontaneous bleed rate per year | 0.6 [0.27 to 1.53]

4. Primary Outcome: Expansion Part: Annualized Bleeding Rate (ABR) for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A "joint bleed" is defined as a bleed with type reported as "joint" and with at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline. A "treated joint bleed" is a joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Treated bleeds that fulfilled the 72-hour rule were included in the analysis of joint bleeds, excluding bleeds due to surgery/procedure.
Time Frame: From Baseline to at least 24 weeks
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Number (95% Confidence Interval); unit: treated joint bleed rate per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
treated joint bleed rate per year | 1.7 [0.82 to 3.68]

5. Primary Outcome: Expansion Part: Annualized Bleeding Rate (ABR) for Treated Target Joint Bleeds
Description: The number of treated target joint bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A "target joint bleed" is defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry. A "treated target joint bleed" is a target joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to at least 24 weeks
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Number (95% Confidence Interval); unit: treated target joint bleed rate per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
treated target joint bleed rate per year | 1.0 [0.31 to 3.26]

6. Secondary Outcome: Expansion Part: Change From Baseline to Week 25 in the Hemophilia A Quality of Life (Haem-A-QoL) Questionnaire Total Score for Adult Participants (≥18 Years of Age)
Description: The Haem-A-QoL is a patient-reported questionnaire that was designed for adult participants with hemophilia. It consists of 46 items comprising 10 dimensions (physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feelings, relationships, treatment, view of yourself, and outlook for the future) and a scale representing Total Score. Items are rated along five response options: never, rarely, sometimes, often, or all the time; although for some items there is also a "not applicable" option. Scale scores range from 0 to 100 with lower scores reflective of better quality of life. A decrease of 7 points or more on the Total Score was defined as the threshold for a clinically meaningful improvement.
Time Frame: Baseline, Week 25
Population: The analysis included all adult participants enrolled in the expansion part of the study. The number analyzed represents participants who completed the questionnaire at Baseline and Week 25.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 37
units on a scale | -13.62 [-18.36 to -8.88]

7. Secondary Outcome: Expansion Part: Percentage of Adult Participants (≥18 Years of Age) With a Clinically Meaningful Improvement From Baseline to Week 25 in the Haem-A-QoL Questionnaire Total Score
Description: as for outcome 6
Time Frame: Baseline, Week 25
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 37
percentage of participants | 67.6

8. Secondary Outcome: Expansion Part: Change From Baseline to Week 25 in the Haem-A-QoL Questionnaire Physical Health Score for Adult Participants (≥18 Years of Age)
Description: The Haem-A-QoL is a patient-reported questionnaire that was designed for adult participants with hemophilia. It consists of 46 items comprising 10 dimensions (physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feelings, relationships, treatment, view of yourself, and outlook for the future) and a scale representing Total Score. Items are rated along five response options: never, rarely, sometimes, often, or all the time; although for some items there is also a "not applicable" option. Scale scores range from 0 to 100 with lower scores reflective of better quality of life. A decrease of 10 points or more on the Physical Health Score was defined as the threshold for a clinically meaningful improvement.
Time Frame: Baseline, Week 25
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 37
units on a scale | -15.14 [-22.44 to -7.83]

9. Secondary Outcome: Expansion Part: Percentage of Adult Participants (≥18 Years of Age) With a Clinically Meaningful Improvement From Baseline to Week 25 in the Haem-A-QoL Questionnaire Physical Health Score
Description: as for outcome 8
Time Frame: Baseline, Week 25
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 37
percentage of participants | 67.6

10. Secondary Outcome: Expansion Part: Change From Baseline to Week 25 in the Hemophilia-Quality of Life-Short Form (Haemo-QoL-SF) Questionnaire Total Score for Adolescent Participants (12-17 Years of Age)
Description: The Haemo-QoL-SF was developed in a series of age-related questionnaires to measure health-related quality of life (HRQoL) in children and adolescents with hemophilia. The short version for older children containing 35 items was selected for adolescents in this study. Items are rated along five response options: never, rarely, sometimes, often, or all the time. This version covers nine dimensions considered relevant for the children's HRQoL (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia, and treatment). Scale scores range from 0 to 100, with lower scores indicating better HRQoL. Given the small number of adolescent participants, the results of the Haemo-QoL-SF questionnaire should be interpreted with caution.
Time Frame: Baseline, Week 25
Population: The analysis included all adolescent participants enrolled in the expansion part of the study. The number analyzed represents participants who completed the questionnaire at Baseline and Week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 3
units on a scale | -8.10 (6.48)

11. Secondary Outcome: Expansion Part: Change From Baseline to Week 25 in the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Questionnaire Visual Analogue Scale (VAS) Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. An increase in the VAS score of 7 points or greater was defined as the threshold for a meaningful improvement.
Time Frame: Baseline, Week 25
Population: The analysis included all participants enrolled in the expansion part of the study. The number analyzed represents participants who completed the questionnaire at Baseline and Week 25.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 40
units on a scale | 5.53 [1.15 to 9.90]

12. Secondary Outcome: Expansion Part: Percentage of Participants With a Meaningful Improvement From Baseline to Week 25 in the EQ-5D-5L Questionnaire VAS Score
Description: as for outcome 11
Time Frame: Baseline, Week 25
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 40
percentage of participants | 35.0

13. Secondary Outcome: Expansion Part: Change From Baseline to Week 25 in the EQ-5D-5L Questionnaire Index Utility Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Published weighting systems allow for creation of a single summary score for the Index Utility Score where overall scores range from 0 to 1, with lower scores representing a higher level of dysfunction. An increase in the Index Utility Score of 0.07 points or greater was defined as the threshold for a meaningful improvement.
Time Frame: Baseline, Week 25
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 40
units on a scale | 0.06 [0.03 to 0.10]

14. Secondary Outcome: Expansion Part: Percentage of Participants With a Meaningful Improvement From Baseline to Week 25 in the EQ-5D-5L Questionnaire Index Utility Score
Description: as for outcome 13
Time Frame: Baseline, Week 25
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 40
percentage of participants | 47.5

15. Secondary Outcome: Expansion Part: Proportion of Days Away From Work to Expected Days at Work in the Previous Four Weeks
Description: Participants enrolled in the expansion part of the study reported at each time point the number of days away from work (i.e., days of work missed) and the expected number of days at work in the previous four weeks, which is reported here for each time point as the proportion of the number of days away from work to the expected number of days at work.
Time Frame: Predose at Baseline, Weeks 13 and 25
Population: The analysis included all participants enrolled in the expansion part of the study who were working and completed the questionnaire at Baseline, Week 13, and Week 25.
Measure: Mean (95% Confidence Interval); unit: away/expected work days
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 28
away/expected work days
  Baseline | 0.05 [0.01 to 0.10]
  Week 13 | 0.00 [0.00 to 0.00]
  Week 25: number analyzed (Participants) | 27
  Week 25 | 0.01 [0.00 to 0.02]

16. Secondary Outcome: Expansion Part: Proportion of Days Away From School to Expected Days at School in the Previous Four Weeks
Description: Participants enrolled in the expansion part of the study reported at each time point the number of days away from school (i.e., days of school missed) and the expected number of days at school in the previous four weeks, which is reported here as the proportion of the number of days away from school to the expected number of days at school.
Time Frame: Predose at Baseline, Weeks 13 and 25
Population: The analysis included all participants enrolled in the expansion part of the study who were enrolled in school and completed the questionnaire at Baseline, Week 13, and Week 25.
Measure: Mean (95% Confidence Interval); unit: away/expected school days
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 10
away/expected school days
  Baseline | 0.12 [0.01 to 0.24]
  Week 13: number analyzed (Participants) | 8
  Week 13 | 0.00 [0.00 to 0.00]
  Week 25 | 0.03 [0.00 to 0.10]

17. Secondary Outcome: Expansion Part: Number of Days Hospitalized
Time Frame: From Baseline until at least 24 weeks of treatment (median [min-max] observation time: 25.57 [24.1-29.4] weeks)
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 41
days | 0 (0)

18. Secondary Outcome: Expansion Part: Percentage of Participants Who Preferred Either the New Emicizumab Subcutaneous (SC) Treatment or Their Previous Hemophilia Intravenous (IV) Treatment, or Had No Preference, as Assessed Using the Emicizumab Preference Survey
Description: The Emicizumab Preference Survey is a fit-for-purpose questionnaire developed by the sponsor to record the participant's preference for treatment with intravenous (IV) factor VIIII (FVIII) or subcutaneous (SC) emicizumab, or no preference.
Time Frame: Predose at Week 17
Population: The analysis included all participants enrolled in the expansion part of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 41
percentage of participants
  Prefer the New Emicizumab SC Treatment | 100 [91.40 to 100.00]
  Prefer My Old Hemophilia Treatment (IV) | 0.0 [0.00 to 8.60]
  Have No Preference | 0.0 [0.00 to 8.60]

19. Secondary Outcome: PK Run-In Part: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Emicizumab
Time Frame: Week 1 Day 1 predose (0 hours) and 8 hours postdose, and Week 1 Days 3 and 5, Week 2 Days 8 and 11, Week 3 Days 15 and 18, Week 4 Days 22 and 25, and Day 1 of Weeks 5, 21, 22, 23, 24, and 25
Population: The analysis included all participants enrolled in the PK Run-In part of the study.
Measure: Median (Full Range); unit: day
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
day
  After First Dose (Weeks 1-5) | 6.95 [3.99 to 7.18]
  After Sixth Dose (Weeks 21-25) | 6.98 [6.90 to 14.03]

20. Secondary Outcome: PK Run-In Part: Maximum Observed Plasma Concentration (Cmax) of Emicizumab
Time Frame: as for outcome 19
Population: The analysis included all participants enrolled in the PK Run-In part of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
μg/mL
  After First Dose (Weeks 1-5) | 31.8 (19.3)
  After Sixth Dose (Weeks 21-25) | 62.7 (17.3)

21. Secondary Outcome: PK Run-In Part: Area Under the Plasma Concentration-Time Curve From Time Zero to End of Dosing Interval (AUC[0-tau]) of Emicizumab
Time Frame: as for outcome 19
Population: The analysis included all participants enrolled in the PK Run-In part of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
day*μg/mL
  After First Dose (Weeks 1-5) | 663 (19.6)
  After Sixth Dose (Weeks 21-25) | 1420 (20.7)

22. Secondary Outcome: PK Run-In Part: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Emicizumab
Time Frame: as for outcome 19
Population: The analysis included all participants enrolled in the PK Run-In part of the study. t1/2 was not properly estimated after the first dose due to sampling time and dosing schedule; hence, dependent PK parameters, such as AUC[0-inf], could not be estimated after the sixth dose of emicizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
day*μg/mL
  After First Dose (Weeks 1-5) | 1490 (27.2)
  After Sixth Dose (Weeks 21-25): number analyzed (Participants) | 0

23. Secondary Outcome: PK Run-In Part: Apparent Plasma Terminal Half-Life (t1/2) of Emicizumab
Time Frame: as for outcome 19
Population: The analysis included all participants enrolled in the PK Run-In part of the study. t1/2 was not properly estimated after the first dose due to sampling time and dosing schedule; hence, t1/2 could not be determined after the sixth dose of emicizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
day
  After First Dose (Weeks 1-5) | 29.5 (38.5)
  After Sixth Dose (Weeks 21-25): number analyzed (Participants) | 0

24. Secondary Outcome: PK Run-In Part: Apparent Clearance (CL/F) of Emicizumab
Description: Only CL/F is reported after the first dose; the apparent clearance at steady state (CLss/F) is reported after the sixth dose instead. This is because t1/2 was not properly estimated after the first dose due to sampling time and dosing schedule, and dependent PK parameters, such as CL/F, could not be estimated.
Time Frame: as for outcome 19
Population: The analysis included all participants enrolled in the PK Run-In part of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
mL/h
  After First Dose (Weeks 1-5) | 10.7 (23.9)
  After Sixth Dose (Weeks 21-25) | 11.1 (20.8)

25. Secondary Outcome: PK Run-In Part: Plasma Concentration of Emicizumab at Specified Timepoints
Time Frame: Week 1 Day 1 predose and 8 hours postdose, and Week 1 Days 3 and 5, Week 2 Days 8 and 11, Week 3 Days 15 and 18, Week 4 Days 22 and 25, and Day 1 of Weeks 5, 6, 7, 8, 9, 11, 13, 15, 17, 19, 21, 22, 23, 24, and 25, and every 12 weeks thereafter to Week 265
Population: The analysis included all participants enrolled in the PK Run-In part of the study. The number analyzed represents the number of participants with an evaluable sample at a given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Emicizumab: PK Run-In Cohort
Number analyzed (Participants) | 7
μg/mL
  Week 1, Day 1 - Predose | NA (NA) — Concentration could not be estimated because samples were below the lower limit of quantification (BLQ).
  Week 1, Day 1 - 8 hours | 7.0 (71.7)
  Week 1, Day 3 | 20.6 (51.2)
  Week 1, Day 5 | 26.5 (29.7)
  Week 2, Day 8 | 29.4 (25.1)
  Week 2, Day 11 | 27.7 (21.9)
  Week 3, Day 15 | 26.3 (20.5)
  Week 3, Day 18 | 24.1 (21.6)
  Week 4, Day 22 | 22.0 (14.8)
  Week 4, Day 25 | 20.6 (15.6)
  Week 5 | 18.5 (18.2)
  Week 6 | 47.4 (13.8)
  Week 7 | 42.1 (18.3)
  Week 8 | 35.4 (22.5)
  Week 9 | 28.2 (18.6)
  Week 11 | 55.9 (20.4)
  Week 13 | 34.6 (24.1)
  Week 15 | 52.0 (17.0)
  Week 17 | 36.7 (16.1)
  Week 19 | 50.8 (32.6)
  Week 21 | 34.5 (25.1)
  Week 22 | 62.2 (17.5)
  Week 23 | 56.5 (19.0)
  Week 24 | 47.9 (28.7)
  Week 25 | 39.2 (25.3)
  Week 37 | 34.0 (15.8)
  Week 49 | 34.7 (23.2)
  Week 61 | 41.1 (25.9)
  Week 73 | 39.7 (22.8)
  Week 85 | 38.0 (29.2)
  Week 97 | 43.6 (17.1)
  Week 109: number analyzed (Participants) | 5
  Week 109 | 37.7 (13.8)
  Week 121: number analyzed (Participants) | 5
  Week 121 | 39.6 (19.8)
  Week 133: number analyzed (Participants) | 5
  Week 133 | 37.5 (14.2)
  Week 145: number analyzed (Participants) | 5
  Week 145 | 34.8 (13.1)
  Week 157: number analyzed (Participants) | 5
  Week 157 | 35.0 (20.7)
  Week 181: number analyzed (Participants) | 5
  Week 181 | 45.4 (14.6)
  Week 193: number analyzed (Participants) | 5
  Week 193 | 37.9 (21.5)
  Week 205: number analyzed (Participants) | 5
  Week 205 | 45.4 (21.0)
  Week 217: number analyzed (Participants) | 5
  Week 217 | 45.3 (11.3)
  Week 229: number analyzed (Participants) | 5
  Week 229 | 52.1 (18.6)
  Week 241: number analyzed (Participants) | 5
  Week 241 | 45.6 (13.6)
  Week 253: number analyzed (Participants) | 5
  Week 253 | 40.4 (13.8)
  Week 265: number analyzed (Participants) | 5
  Week 265 | 42.4 (16.5)

26. Secondary Outcome: Expansion Part: Plasma Concentration of Emicizumab at Specified Timepoints
Time Frame: Predose at Weeks 1, 2, 3, 4, 5, 9, 13, 17, 21, 25, 37, 49, 61, 73. 85, 97, 109, 121, 133, 145, 157, 169, 181, 193, 205, 217, 229, 241, and 253
Population: The analysis included all participants enrolled in the Expansion part of the study. The number analyzed represents the number of participants with an evaluable sample at a given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
μg/mL
  Week 1: number analyzed (Participants) | 40
  Week 1 | NA (NA) — Concentration could not be estimated because samples were below the lower limit of quantification (BLQ).
  Week 2 | 16.0 (36.8)
  Week 3 | 29.8 (30.5)
  Week 4: number analyzed (Participants) | 40
  Week 4 | 41.3 (32.4)
  Week 5 | 48.8 (32.2)
  Week 9 | 40.4 (45.7)
  Week 13: number analyzed (Participants) | 40
  Week 13 | 38.9 (49.1)
  Week 17 | 36.1 (53.8)
  Week 21 | 37.4 (48.3)
  Week 25 | 37.6 (52.5)
  Week 37: number analyzed (Participants) | 38
  Week 37 | 39.6 (49.9)
  Week 49: number analyzed (Participants) | 38
  Week 49 | 40.2 (48.4)
  Week 61: number analyzed (Participants) | 37
  Week 61 | 38.7 (51.7)
  Week 73: number analyzed (Participants) | 34
  Week 73 | 42.1 (51.2)
  Week 85: number analyzed (Participants) | 26
  Week 85 | 36.4 (50.8)
  Week 97: number analyzed (Participants) | 21
  Week 97 | 35.6 (49.5)
  Week 109: number analyzed (Participants) | 20
  Week 109 | 33.0 (63.6)
  Week 121: number analyzed (Participants) | 21
  Week 121 | 32.5 (60.5)
  Week 133: number analyzed (Participants) | 21
  Week 133 | 33.7 (49.0)
  Week 145: number analyzed (Participants) | 14
  Week 145 | 36.5 (51.7)
  Week 157: number analyzed (Participants) | 15
  Week 157 | 47.3 (36.0)
  Week 169: number analyzed (Participants) | 18
  Week 169 | 41.7 (41.9)
  Week 181: number analyzed (Participants) | 15
  Week 181 | 45.1 (47.9)
  Week 193: number analyzed (Participants) | 15
  Week 193 | 48.6 (47.0)
  Week 205: number analyzed (Participants) | 16
  Week 205 | 46.0 (48.2)
  Week 217: number analyzed (Participants) | 15
  Week 217 | 43.9 (47.8)
  Week 229: number analyzed (Participants) | 14
  Week 229 | 50.2 (43.1)
  Week 241: number analyzed (Participants) | 9
  Week 241 | 36.2 (46.5)
  Week 253: number analyzed (Participants) | 9
  Week 253 | 38.8 (46.6)

27. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: The number of participants experiencing at least one adverse event (AE), including all non-serious and serious AEs, is reported here. According to the ICH guideline for Good Clinical Practice, an AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. The terms "severe" and "serious" are not synonymous. A serious AE is any AE that is a significant medical event meeting any of the standard criteria. Severity refers to the intensity of an AE (e.g., rated as mild, moderate, or severe, or according to the World Health Organization [WHO] toxicity grading scale); the event itself may be of relatively minor medical significance. Severity and seriousness were independently assessed by the investigator for each reported AE.
Time Frame: From Baseline to study completion, dose up-titration, or change of dosing regimen, whichever occurred first (up to 5 years, 5 months)
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants
  Any Adverse Event (AE) | 7 | 39
  Serious AE | 2 | 8

28. Secondary Outcome: Number of Participants With at Least One Grade ≥3 Adverse Event
Description: The World Health Organization (WHO) Toxicity Grading Scale was used for assessing adverse event (AE) severity. For AEs that are not specifically listed in the WHO Toxicity Grading Scale, a Grade 3 AE is defined as: severe, marked limitation in activity, some assistance usually required, medical intervention or therapy required, hospitalization possible; and a Grade 4 AE is defined as: life-threatening, extreme limitation in activity, significant assistance required, significant medical intervention or therapy required, hospitalization or hospice care probable. The terms "severe" and "serious" are not synonymous. A serious AE is any AE that is a significant medical event meeting any of the standard criteria. Severity refers to the intensity of an AE; the event itself may be of relatively minor medical significance. Severity and seriousness were independently assessed by the investigator for each reported AE.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 2 | 7

29. Secondary Outcome: Number of Participants With at Least One Adverse Event Leading to Withdrawal From Treatment
Description: According to the ICH guideline for Good Clinical Practice, an AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. The terms "severe" and "serious" are not synonymous. A serious AE is any AE that is a significant medical event meeting any of the standard criteria. Severity refers to the intensity of an AE (e.g., rated as mild, moderate, or severe, or according to the World Health Organization [WHO] toxicity grading scale); the event itself may be of relatively minor medical significance. Severity and seriousness were independently assessed by the investigator for each reported AE.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 0 | 0

30. Secondary Outcome: Number of Participants With at Least One Adverse Event Related to Study Treatment
Description: According to the ICH guideline for Good Clinical Practice, an adverse event (AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. In order to assess the causality of an AE, investigators used their knowledge of the patient, the circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether an AE is considered to be related to the study drug, indicating "yes" or "no" accordingly.
Time Frame: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants
  Any Adverse Event Related to Study Treatment | 2 | 14
  Injection Site Reaction | 1 | 9
  Chills | 0 | 1
  Presyncope | 0 | 1
  Rash | 0 | 1
  Erythema | 0 | 1
  Incorrect Dose Administered | 0 | 1
  Accidental Overdose | 0 | 1
  Iron Deficiency Anaemia | 1 | 0

31. Secondary Outcome: Number of Participants With at Least One Adverse Event of Changes From Baseline in Vital Signs
Description: The number of participants with adverse events of changes from baseline in vital signs is reported here. Vital signs measurements consisted of heart and respiratory rate, temperature, and systolic and diastolic blood pressures, with an abnormal vital sign value being outside of the normal range. An abnormal vital sign result was reported as an adverse event if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment (e.g., dosage modification, treatment interruption or discontinuation); resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. All of the adverse events reported here were assessed independently by the investigator as not related to treatment with emicizumab.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants
  Hypertension | 2 | 4
  Pyrexia | 1 | 4
  Tachycardia | 0 | 1

32. Secondary Outcome: Number of Participants With at Least One Adverse Event of Changes From Baseline in Physical Examination Findings
Description: Post-baseline physical examination abnormalities that were not present at baseline or worsened were reported as adverse events.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 0 | 0

33. Secondary Outcome: Number of Participants With at Least One Shift in Clinical Laboratory Parameters From Baseline World Health Organization (WHO) Toxicity Scale Grade 0-2 to Post-Baseline WHO Grade 3 or 4
Description: An abnormal laboratory value was defined as a laboratory test result outside of the normal range for hematology or serum chemistry parameters. The WHO toxicity grading scale, which ranges from Grades 1 to 4 (least severe to most severe, respectively; Grade 0 is within normal range), was used for assessing the severity of laboratory abnormalities and adverse events (WHO 2003). Not every laboratory abnormality qualified as an adverse event; an abnormality was reported as an adverse event if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment (e.g., dosage modification, treatment interruption or discontinuation); resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. In this study, any laboratory value changes were transient and returned to baseline for all participants.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants
  Aspartate Aminotransferase (AST) - High | 0 | 1
  Calcium, Corrected - Low | 0 | 1
  Phosphorus - Low | 0 | 2
  Sodium - High | 0 | 1

34. Secondary Outcome: Number of Participants With at Least One Local Injection-Site Reaction
Description: Local adverse events that occurred within 24 hours after study drug administration and, in the investigator's opinion, were judged to be related to study drug injection, were captured as an "injection-site reaction" on the Adverse Event electronic Case Report Form (eCRF). An injection-related reaction that was localized was marked as a "local injection-site reaction."
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 1 | 9

35. Secondary Outcome: Number of Participants With at Least One Thromboembolic Event
Description: Hypercoagulation and thromboembolic events were to be reported as serious adverse events or adverse events of special interest. Healthcare providers educated patients/caregivers to recognize the signs and symptoms of potential thromboembolism (i.e., dyspnea, chest pain, leg pain or swelling, etc.) and to ensure that they understood the importance of seeking appropriate medical attention.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 0 | 0

36. Secondary Outcome: Number of Participants With at Least One Thrombotic Microangiopathy
Description: Thrombotic microangiopathy is used to describe a group of disorders with clinical features of microangiopathic hemolytic anemia, thrombocytopenia, and organ damage that can include the kidneys, gastrointestinal system, or central nervous system, etc. Thrombotic microangiopathy events were to be reported as serious adverse events or adverse events of special interest.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 0 | 0

37. Secondary Outcome: Number of Participants With at Least One Systemic Hypersensitivity, Anaphylaxis, or Anaphylactoid Reaction
Description: Since emicizumab is a biological product, acute, systemic hypersensitivity reactions, including anaphylaxis and anaphylactic reactions, may occur. These events were to be reported as serious adverse events or adverse events of special interest. Healthcare providers (HCP) instructed patients and caregivers how to recognize the signs and symptoms of hypersensitivity, anaphylactic, and anaphylactoid reactions and to contact an HCP or seek emergency care in case of any such occurrence.
Time Frame: as for outcome 27
Population: The analysis included all participants who received at least one dose of emicizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 0 | 0

38. Secondary Outcome: Number of Participants With Anti-Drug Antibodies to Emicizumab at Any Time Post-Baseline During the Study
Description: A validated enzyme-linked immunosorbent assay (ELISA) method was used to analyze the levels of anti-drug antibodies (ADAs) to emicizumab in blood plasma samples. Participants were considered ADA-positive if they were ADA-negative at baseline but developed an ADA response following study drug administration (treatment-induced ADA response), or if they were ADA-positive at baseline and the titer of one or more post-baseline samples was at least 4-fold greater (i.e., ≥ 0.60 titer units) than the titer of the baseline sample (treatment-enhanced ADA response).
Time Frame: Baseline, Weeks 5, 9, 13, 17, 21, and 25, and every 12 weeks thereafter until study completion (up to 5 years, 5 months)
Population: The analysis included all participants who received at least one dose of emicizumab. The number analyzed indicates those with both baseline and post-baseline assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 7 | 41
Participants | 1 | 1

39. Secondary Outcome: Number of Participants With De Novo Development of Anti-Factor VIII (FVIII) Antibodies
Description: The levels of anti-FVIII antibodies (inhibitors) were analyzed using a validated FVIII activity assay. A participant was considered to have developed de novo FVIII inhibitors if the inhibitor levels detected in a post-baseline sample reached or exceeded a pre-determined threshold.
Time Frame: Baseline, Weeks 9 and 17 (for non-inhibitor subjects only), Week 25, and every 12 weeks thereafter until study completion (up to 5 years, 5 months)
Population: The analysis included all participants who were FVIII inhibitor-negative at baseline and had received at least one dose of emicizumab during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 4 | 36
Participants | 0 | 0

40. Secondary Outcome: Long-Term Efficacy of Emicizumab: Model-Based Annualized Bleeding Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds
Description: The number of bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (≥) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration or change of dosing regimen were excluded.
Time Frame: From start of emicizumab treatment to study completion, dose up-titration, or change of dosing regimen (median [min-max] efficacy period for all emicizumab participants: 191.14 [28.0-264.4] weeks)
Population: The analysis includes all participants in the Expansion Cohort who received emicizumab on the study.
Measure: Number (95% Confidence Interval); unit: bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
bleeds per year
  Treated Bleeds | 1.9 [1.22 to 3.02]
  All Bleeds | 2.9 [1.97 to 4.17]
  Treated Spontaneous Bleeds | 0.5 [0.26 to 1.00]
  Treated Joint Bleeds | 1.2 [0.69 to 2.17]
  Treated Target Joint Bleeds | 0.5 [0.24 to 1.26]

41. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds
Description: The number of bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (≥) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration or change of dosing regimen were excluded.
Time Frame: as for outcome 40
Population: The analysis includes all participants in the Expansion Cohort who received emicizumab on the study.
Measure: Mean (95% Confidence Interval); unit: bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
bleeds per year
  Treated Bleeds | 2.0 [0.25 to 7.28]
  All Bleeds | 3.0 [0.63 to 8.82]
  Treated Spontaneous Bleeds | 0.7 [0.00 to 4.95]
  Treated Joint Bleeds | 1.3 [0.07 to 6.11]
  Treated Target Joint Bleeds | 0.6 [0.00 to 4.77]

42. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds
Description: as for outcome 41
Time Frame: as for outcome 40
Population: The analysis includes all participants in the Expansion Cohort who received emicizumab on the study.
Measure: Median (Inter-Quartile Range); unit: bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
bleeds per year
  Treated Bleeds | 0.6 [0.20 to 2.20]
  All Bleeds | 1.2 [0.60 to 3.78]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 0.59]
  Treated Joint Bleeds | 0.3 [0.00 to 1.22]
  Treated Target Joint Bleeds | 0.0 [0.00 to 0.20]

43. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds Per 12-Week Intervals Over Time
Description: The number of treated bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: a bleed for which coagulation factors were administered. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants with dose up-titration or a change in emicizumab dosing regimen (after implementation of protocol v5), the efficacy period ended the day before the first day on the up-titrated dose or changed dosing regimen.
Time Frame: 1-12, 13-24, 25-36, 37-48, 49-60, 61-72, 73-84, 85-96, 97-108, 109-120, 121-132, 133-144, 145-156, 157-168, 169-180, 181-192, 193-204, 205-216, 217-228, 229-240, 241-252, and 253-264 weeks
Population: The analysis includes all participants in the Expansion Cohort who received emicizumab on the study. The number analyzed includes participants with available data over each interval.
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
Treated bleeds per year
  1 to 12 Weeks | 2.3 [0.35 to 7.75]
  13 to 24 Weeks | 2.5 [0.43 to 8.08]
  25 to 36 Weeks: number analyzed (Participants) | 38
  25 to 36 Weeks | 1.5 [0.11 to 6.40]
  37 to 48 Weeks: number analyzed (Participants) | 38
  37 to 48 Weeks | 1.9 [0.23 to 7.14]
  49 to 60 Weeks: number analyzed (Participants) | 38
  49 to 60 Weeks | 1.3 [0.06 to 6.01]
  61 to 72 Weeks: number analyzed (Participants) | 36
  61 to 72 Weeks | 2.7 [0.48 to 8.25]
  73 to 84 Weeks: number analyzed (Participants) | 32
  73 to 84 Weeks | 1.1 [0.04 to 5.72]
  85 to 96 Weeks: number analyzed (Participants) | 24
  85 to 96 Weeks | 1.4 [0.10 to 6.33]
  97 to 108 Weeks: number analyzed (Participants) | 22
  97 to 108 Weeks | 2.0 [0.23 to 7.19]
  109 to 120 Weeks: number analyzed (Participants) | 22
  109 to 120 Weeks | 1.4 [0.08 to 6.22]
  121 to 132 Weeks: number analyzed (Participants) | 22
  121 to 132 Weeks | 1.8 [0.18 to 6.87]
  133 to 144 Weeks: number analyzed (Participants) | 22
  133 to 144 Weeks | 1.0 [0.02 to 5.55]
  145 to 156 Weeks: number analyzed (Participants) | 22
  145 to 156 Weeks | 1.6 [0.13 to 6.55]
  157 to 168 Weeks: number analyzed (Participants) | 22
  157 to 168 Weeks | 2.0 [0.23 to 7.19]
  169 to 180 Weeks: number analyzed (Participants) | 21
  169 to 180 Weeks | 2.1 [0.26 to 7.34]
  181 to 192 Weeks: number analyzed (Participants) | 20
  181 to 192 Weeks | 1.3 [0.07 to 6.09]
  193 to 204 Weeks: number analyzed (Participants) | 18
  193 to 204 Weeks | 1.7 [0.15 to 6.73]
  205 to 216 Weeks: number analyzed (Participants) | 18
  205 to 216 Weeks | 1.4 [0.10 to 6.33]
  217 to 228 Weeks: number analyzed (Participants) | 18
  217 to 228 Weeks | 1.2 [0.05 to 5.93]
  229 to 240 Weeks: number analyzed (Participants) | 18
  229 to 240 Weeks | 1.0 [0.02 to 5.51]
  241 to 252 Weeks: number analyzed (Participants) | 16
  241 to 252 Weeks | 2.4 [0.40 to 7.92]
  253 to 264 Weeks: number analyzed (Participants) | 5
  253 to 264 Weeks | 2.6 [0.46 to 8.17]

44. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds Per 12-Week Intervals Over Time
Description: as for outcome 43
Time Frame: as for outcome 43
Population: as for outcome 43
Measure: Median (Inter-Quartile Range); unit: Treated bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
Treated bleeds per year
  1 to 12 Weeks | 0.0 [0.00 to 4.35]
  13 to 24 Weeks | 0.0 [0.00 to 4.35]
  25 to 36 Weeks: number analyzed (Participants) | 38
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 38
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 38
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 36
  61 to 72 Weeks | 0.0 [0.00 to 2.17]
  73 to 84 Weeks: number analyzed (Participants) | 32
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 24
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 22
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 22
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 22
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 22
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 22
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 22
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 21
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 20
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 18
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 18
  205 to 216 Weeks | 0.0 [0.00 to 4.35]
  217 to 228 Weeks: number analyzed (Participants) | 18
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 18
  229 to 240 Weeks | 0.0 [0.00 to 0.00]
  241 to 252 Weeks: number analyzed (Participants) | 16
  241 to 252 Weeks | 0.0 [0.00 to 4.35]
  253 to 264 Weeks: number analyzed (Participants) | 5
  253 to 264 Weeks | 4.3 [0.00 to 4.35]

45. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for All Bleeds Per 12-Week Intervals Over Time
Description: The number of all bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. All bleeds included both treated bleeds (with coagulation factors) and non-treated bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants with dose up-titration or a change in emicizumab dosing regimen (after implementation of protocol v5), the efficacy period ended the day before the first day on the up-titrated dose or changed dosing regimen.
Time Frame: as for outcome 43
Population: as for outcome 43
Measure: Mean (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
All bleeds per year
  1 to 12 Weeks | 5.1 [1.67 to 11.80]
  13 to 24 Weeks | 4.0 [1.11 to 10.29]
  25 to 36 Weeks: number analyzed (Participants) | 38
  25 to 36 Weeks | 3.1 [0.66 to 8.90]
  37 to 48 Weeks: number analyzed (Participants) | 38
  37 to 48 Weeks | 2.5 [0.42 to 8.03]
  49 to 60 Weeks: number analyzed (Participants) | 38
  49 to 60 Weeks | 2.2 [0.30 to 7.50]
  61 to 72 Weeks: number analyzed (Participants) | 36
  61 to 72 Weeks | 3.5 [0.85 to 9.52]
  73 to 84 Weeks: number analyzed (Participants) | 32
  73 to 84 Weeks | 1.8 [0.17 to 6.85]
  85 to 96 Weeks: number analyzed (Participants) | 24
  85 to 96 Weeks | 2.0 [0.24 to 7.21]
  97 to 108 Weeks: number analyzed (Participants) | 22
  97 to 108 Weeks | 2.4 [0.37 to 7.81]
  109 to 120 Weeks: number analyzed (Participants) | 22
  109 to 120 Weeks | 1.6 [0.13 to 6.55]
  121 to 132 Weeks: number analyzed (Participants) | 22
  121 to 132 Weeks | 2.2 [0.30 to 7.50]
  133 to 144 Weeks: number analyzed (Participants) | 22
  133 to 144 Weeks | 1.2 [0.05 to 5.89]
  145 to 156 Weeks: number analyzed (Participants) | 22
  145 to 156 Weeks | 2.0 [0.23 to 7.19]
  157 to 168 Weeks: number analyzed (Participants) | 22
  157 to 168 Weeks | 2.0 [0.23 to 7.19]
  169 to 180 Weeks: number analyzed (Participants) | 21
  169 to 180 Weeks | 2.3 [0.33 to 7.66]
  181 to 192 Weeks: number analyzed (Participants) | 20
  181 to 192 Weeks | 1.7 [0.17 to 6.81]
  193 to 204 Weeks: number analyzed (Participants) | 18
  193 to 204 Weeks | 1.9 [0.22 to 7.12]
  205 to 216 Weeks: number analyzed (Participants) | 18
  205 to 216 Weeks | 1.4 [0.10 to 6.33]
  217 to 228 Weeks: number analyzed (Participants) | 18
  217 to 228 Weeks | 1.7 [0.15 to 6.73]
  229 to 240 Weeks: number analyzed (Participants) | 18
  229 to 240 Weeks | 1.0 [0.02 to 5.51]
  241 to 252 Weeks: number analyzed (Participants) | 16
  241 to 252 Weeks | 2.4 [0.40 to 7.92]
  253 to 264 Weeks: number analyzed (Participants) | 5
  253 to 264 Weeks | 2.6 [0.46 to 8.17]

46. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for All Bleeds Per 12-Week Intervals Over Time
Description: as for outcome 45
Time Frame: as for outcome 43
Population: as for outcome 43
Measure: Median (Inter-Quartile Range); unit: All bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
All bleeds per year
  1 to 12 Weeks | 0.0 [0.00 to 8.70]
  13 to 24 Weeks | 4.3 [0.00 to 4.35]
  25 to 36 Weeks: number analyzed (Participants) | 38
  25 to 36 Weeks | 0.0 [0.00 to 4.35]
  37 to 48 Weeks: number analyzed (Participants) | 38
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 38
  49 to 60 Weeks | 0.0 [0.00 to 4.35]
  61 to 72 Weeks: number analyzed (Participants) | 36
  61 to 72 Weeks | 0.0 [0.00 to 4.35]
  73 to 84 Weeks: number analyzed (Participants) | 32
  73 to 84 Weeks | 0.0 [0.00 to 4.35]
  85 to 96 Weeks: number analyzed (Participants) | 24
  85 to 96 Weeks | 0.0 [0.00 to 2.17]
  97 to 108 Weeks: number analyzed (Participants) | 22
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 22
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 22
  121 to 132 Weeks | 0.0 [0.00 to 4.35]
  133 to 144 Weeks: number analyzed (Participants) | 22
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 22
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 22
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 21
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 20
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 18
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 18
  205 to 216 Weeks | 0.0 [0.00 to 4.35]
  217 to 228 Weeks: number analyzed (Participants) | 18
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 18
  229 to 240 Weeks | 0.0 [0.00 to 0.00]
  241 to 252 Weeks: number analyzed (Participants) | 16
  241 to 252 Weeks | 0.0 [0.00 to 4.35]
  253 to 264 Weeks: number analyzed (Participants) | 5
  253 to 264 Weeks | 4.3 [0.00 to 4.35]

47. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for Treated Spontaneous Bleeds Per 12-Week Intervals Over Time
Description: The number of treated spontaneous bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated spontaneous bleeds were defined as treated (with coagulation factors) bleeds with no known contributing factor (e.g., trauma, surgery). The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants with dose up-titration or a change in emicizumab dosing regimen (after implementation of protocol v5), the efficacy period ended the day before the first day on the up-titrated dose or changed dosing regimen.
Time Frame: as for outcome 43
Population: as for outcome 43
Measure: Mean (95% Confidence Interval); unit: Treated spontaneous bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
Treated spontaneous bleeds per year
  1 to 12 Weeks | 0.4 [0.00 to 4.35]
  13 to 24 Weeks | 1.0 [0.02 to 5.49]
  25 to 36 Weeks: number analyzed (Participants) | 38
  25 to 36 Weeks | 0.1 [0.00 to 3.93]
  37 to 48 Weeks: number analyzed (Participants) | 38
  37 to 48 Weeks | 0.0 [0 to 3.69]
  49 to 60 Weeks: number analyzed (Participants) | 38
  49 to 60 Weeks | 0.3 [0.00 to 4.38]
  61 to 72 Weeks: number analyzed (Participants) | 36
  61 to 72 Weeks | 0.2 [0.00 to 4.18]
  73 to 84 Weeks: number analyzed (Participants) | 32
  73 to 84 Weeks | 0.1 [0.00 to 3.97]
  85 to 96 Weeks: number analyzed (Participants) | 24
  85 to 96 Weeks | 0.0 [0 to 3.69]
  97 to 108 Weeks: number analyzed (Participants) | 22
  97 to 108 Weeks | 0.2 [0.00 to 4.09]
  109 to 120 Weeks: number analyzed (Participants) | 22
  109 to 120 Weeks | 0.4 [0.00 to 4.48]
  121 to 132 Weeks: number analyzed (Participants) | 22
  121 to 132 Weeks | 0.4 [0.00 to 4.48]
  133 to 144 Weeks: number analyzed (Participants) | 22
  133 to 144 Weeks | 0.4 [0.00 to 4.48]
  145 to 156 Weeks: number analyzed (Participants) | 22
  145 to 156 Weeks | 1.0 [0.02 to 5.55]
  157 to 168 Weeks: number analyzed (Participants) | 22
  157 to 168 Weeks | 1.8 [0.18 to 6.87]
  169 to 180 Weeks: number analyzed (Participants) | 21
  169 to 180 Weeks | 0.0 [0 to 3.69]
  181 to 192 Weeks: number analyzed (Participants) | 20
  181 to 192 Weeks | 0.0 [0 to 3.69]
  193 to 204 Weeks: number analyzed (Participants) | 18
  193 to 204 Weeks | 0.7 [0.01 to 5.09]
  205 to 216 Weeks: number analyzed (Participants) | 18
  205 to 216 Weeks | 0.5 [0.00 to 4.64]
  217 to 228 Weeks: number analyzed (Participants) | 18
  217 to 228 Weeks | 0.0 [0 to 3.69]
  229 to 240 Weeks: number analyzed (Participants) | 18
  229 to 240 Weeks | 0.2 [0.00 to 4.18]
  241 to 252 Weeks: number analyzed (Participants) | 16
  241 to 252 Weeks | 0.8 [0.01 to 5.25]
  253 to 264 Weeks: number analyzed (Participants) | 5
  253 to 264 Weeks | 0.0 [0 to 3.69]

48. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for Treated Spontaneous Bleeds Per 12-Week Intervals Over Time
Description: as for outcome 47
Time Frame: as for outcome 43
Population: as for outcome 43
Measure: Median (Inter-Quartile Range); unit: Treated spontaneous bleeds per year
Arm/Group | Emicizumab: Expansion Cohort
Number analyzed (Participants) | 41
Treated spontaneous bleeds per year
  1 to 12 Weeks | 0.0 [0.00 to 0.00]
  13 to 24 Weeks | 0.0 [0.00 to 0.00]
  25 to 36 Weeks: number analyzed (Participants) | 38
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 38
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 38
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 36
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 32
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 24
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 22
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 22
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 22
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 22
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 22
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 22
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 21
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 20
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 18
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 18
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 18
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 18
  229 to 240 Weeks | 0.0 [0.00 to 0.00]
  241 to 252 Weeks: number analyzed (Participants) | 16
  241 to 252 Weeks | 0.0 [0.00 to 0.00]
  253 to 264 Weeks: number analyzed (Participants) | 5
  253 to 264 Weeks | 0.0 [0.00 to 0.00]

ADVERSE EVENTS:
Time Frame: From Baseline to study completion, dose up-titration, or change of dosing regimen, whichever occurred first (up to 5 years, 5 months)
Arm/Group | Emicizumab: PK Run-In Cohort | Emicizumab: Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/7 | 8/41
Other Adverse Events (participants affected / at risk) | 7/7 | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emicizumab: PK Run-In Cohort (N=7) | Emicizumab: Expansion Cohort (N=41)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS OBSTRUCTIVE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR COMPRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DEVICE LOOSENING (Product Issues) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emicizumab: PK Run-In Cohort (N=7) | Emicizumab: Expansion Cohort (N=41)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ECZEMA EYELIDS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (3)
DYSPEPSIA (Gastrointestinal disorders) | 1 (3) | 0 (0)
ODYNOPHAGIA (Gastrointestinal disorders) | 2 (3) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 5 (5)
CHEST PAIN (General disorders) | 1 (2) | 1 (1)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 (1) | 0 (0)
INFLAMMATION (General disorders) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 1 (1) | 9 (40)
MEDICAL DEVICE DISCOMFORT (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 3 (4)
PYREXIA (General disorders) | 1 (1) | 4 (5)
SEASONAL ALLERGY (Immune system disorders) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 6 (6)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (3) | 0 (0)
EAR INFECTION (Infections and infestations) | 2 (2) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 14 (17)
PHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TINEA CAPITIS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 3 (5)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
GINGIVAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 3 (5)
POST PROCEDURAL INFLAMMATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TONGUE INJURY (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (18) | 17 (43)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (7) | 6 (8)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GREATER TROCHANTERIC PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT LOCK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (8)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (5)
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (7) | 12 (17)
MOTOR DYSFUNCTION (Nervous system disorders) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1)
DEVICE BREAKAGE (Product Issues) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
HYPERTENSION (Vascular disorders) | 2 (2) | 4 (7)

LIMITATIONS AND CAVEATS:
Given the small number of adolescent participants, the results of the Haemo-QoL-SF questionnaire should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03020160/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03020160/SAP_001.pdf